CLINICAL TRIAL: NCT04947085
Title: Comparison of Nebulized Ketamine to Intravenous Sub-Dissociative Dose Ketamine for Treating Acute and Chronic Painful Conditions in the ED: A Prospective, Randomized, Double-Blind, Double-Dummy Clinical Trial.
Brief Title: Comparison of Nebulized Ketamine to Intravenous Sub-Dissociative Dose Ketamine for Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Antonios Likourezos (Other)
Responsible Party: Sponsor-Investigator, Antonios Likourezos, Research Administration Director, Maimonides Medical Center
Organization: Maimonides Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020-08-05
Record Dates: First submitted 2021-06-23; First posted 2021-07-01 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2023-11

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- IV SDK (Active Comparator): intravenous ketamine administration in sub-dissociative doses (SDK) administered at 0.3 mg/kg over 15 minutes to patients presenting to the ED of Maimonides Medical Center with acute and chronic painful conditions.
  Interventions: Drug: Ketamine via Intravenous
- K-BAN (Active Comparator): nebulized ketamine at 0.75mg/kg administered via BAN to patients presenting to the ED of Maimonides Medical Center with acute and chronic painful conditions.
  Interventions: Drug: Ketamine via BAN

INTERVENTIONS:
Drug: Ketamine via Intravenous — Ketamine administration in sub-dissociative doses
  Arms: IV SDK
Drug: Ketamine via BAN — Ketamine administered via Breath-Actuated Nebulizer (BAN)
  Arms: K-BAN

SUMMARY:
Ketamine is a non-competitive N-methyl-D-aspartate (NMDA)/glutamate receptor complex antagonist that decreases pain by diminishing central sensitization, hyperalgesia, and "wind-up" phenomenon at the level of the spinal cord (dorsal ganglion) and central nervous system (1). Ketamine administration in sub-dissociative doses (SDK) of 0.1-0.3 mg/kg in pre-hospital settings and in the ED results in effective pain relief in patients with acute traumatic and non-traumatic pain, chronic non-cancer and cancer pain, and in patients with opioid-tolerant pain by virtue of providing anti-hyperalgesia, anti-allodynia, and anti-tolerance (2-4). Two commonly utilized routes of SDK administration in the ED include an intravenous route (intravenous push dose or short infusion) and intranasal route.

In the situation when intravenous access is not readily available or unobtainable, and intranasal route is not feasible, another non-invasive route of ketamine administration such as inhalation via Breath-Actuated Nebulizer (BAN) is coming into the play. The BAN allows a controlled patient-initiated delivery of analgesics in titratable fashion. Nebulized administration of ketamine has been studied in the areas of acute postoperative pain management (post-intubational sore throat), in anesthesia (pre-medication for general anesthesia,) and in managing cancer pain, and status asthmaticus therapy.

However, our research team has published a case series of 5 patients receiving nebulized ketamine for a variety of acute painful conditions and has recently completed a randomized double-blind trial of 120 adult patients that evaluated analgesic efficacy and safety of nebulized ketamine at three different dosing regimens for acute pain in the ED. Currently, we are conducting two additional studies evaluating the role of nebulized ketamine in pediatric ED and pre-hospital arena.

In this study the investigators hypothesize that intravenous sub-dissociative-dose ketamine of 0.3 mg/kg will provide better analgesia at 30 min post-medication administration in comparison to nebulized ketamine administered at 0.75 mg/kg. The primary outcome of this trial is the comparative reduction in participant's pain scores at 30 minutes post medication administration.

DETAILED DESCRIPTION:
Design: This is a prospective, randomized, double-blind, double dummy trial comparing analgesic efficacy and safety of intravenous SDK administered at 0.3 mg/kg over 15 minutes to nebulized ketamine at 0.75mg/kg administered via BAN to patients presenting to the ED of Maimonides Medical Center with acute and chronic painful conditions. Upon meeting the eligibility criteria, patients will be randomized into two study groups: IV SDK and Nebulized K-BAN.

Subjects: Patients 18 years of age and older presenting to the ED with acute and chronic painful conditions such as traumatic and non-traumatic abdominal, flank, back, musculoskeletal pain, headache, as well as exacerbation of chronic abdominal, musculoskeletal and neuropathic pain with a score of 5 or more on a standard 11- point (0 to 10) numeric rating scale and requiring parenteral analgesia as determined by the treating attending physician. Patients' screening and enrollment will be performed by study investigators and research assistants. All patients will be enrolled at various times of the day when study investigators will be available for patient enrollment and an ED pharmacist will be available for medication preparation

Data Collection Procedures: Each patient will be approached by a study investigator for acquisition of written informed consent and Health Insurance Portability and Accountability Act authorization after being evaluated by the treating emergency physician and determined to meet study eligibility criteria. When English will not be the participant's primary language, a language- appropriate consent form will be used and non-investigator, hospital-employed, trained interpreters or licensed telephone interpreter will assist in acquisition of informed consent. Baseline pain score will be determined with an 11-point numeric rating scale (0 to 10), described to the patient as "no pain" being 0 and "the worst pain imaginable" being 10. A study investigator will record the patient's body weight and baseline vital signs.

The on-duty ED pharmacist will prepare either a breath-actuated nebulizer with a dose of 0.75 mg/kg or an infusion dose of IV SDK at 0.3 mg/kg in 100 ml normal saline bag according to the predetermined randomization list, which will be created in SPSS (version 24; IBM Corp, Armonk, NY) with block randomization of every 10 participants. All participants will receive a corresponding placebo in order to maintain double-dummy design: the subjects randomized to receive IV SDK will also receive nebulized saline via BAN, and the subjects receiving K-BAN will also receive an IV infusion of Normal Saline over 15 minutes. The medication will be delivered to the treating nurse in a blinded fashion who will set up an infusion pump with a run time of 15 minutes. The nebulization of active drug and placebo via BAN will have a minimum time of 5 min and maximum time of 15 min.

Study investigators will record pain scores, vital signs, and adverse effects at 15, 30, 60, 90, and 120 minutes. If patients reported a pain numeric rating scale score of 5 or greater and requested additional pain relief, intravenous morphine at 0.1 mg/kg will be administered as a rescue analgesic.

The preparing ED pharmacist, research manager, and statistician will be the only ones with knowledge of the study arm to which each participant would be randomized. Treating providers, participants, and the data collecting research team will be blind to the medication route received.

All data will be recorded on data collection sheets, including patients' sex, demographics, medical history, and vital signs, and entered into SPSS (version 24.0; IBM Corp) by the research manager. Development of the randomization list, confirmation of written consent acquisition for all participants, and statistical analyses will be conducted by the research administrator and/or statistician who will work independently of any data collection.

Patients will be closely monitored for any change in vital sings and for adverse effects during the entire study period (up to 120 minutes) by study investigators. Common adverse effects that are associated with sub-dissociative dose ketamine are felling of unreality, dizziness, nausea, vomiting, and sedation.

ELIGIBILITY:
Inclusion Criteria:

* ED patients
* Patients 18 years of age
* acute and chronic painful conditions
* pain with a score of 5 or more on a standard 11- point (0 to 10) numeric rating scale.
* Patients will have to be awake, alert, and oriented to person, place, and time,
* Be able to demonstrate understanding of the informed consent process and content.
* Patients also will have to demonstrate ability to verbalize the nature of any adverse effects they might experience as well as to express their pain severity by using the NRS.

Exclusion Criteria:

* Altered mental status,
* allergy to ketamine,
* pregnant patients,
* weight greater than 150 kg,
* unstable vital signs (systolic blood pressure <90 or>180 mm Hg, pulse rate <50 or >150 beats/min, and respiration rate <10 or >30 breaths/min),
* inability to provide consent,
* past medical history of alcohol or drug abuse, or schizophrenia.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Motov, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IV SDK | K-BAN
Started | 75 | 75
Completed | 72 | 75
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IV SDK | K-BAN | Total
Number analyzed (Participants) | 75 | 75 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (13) | 47 (16) | 46.6 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 39 | 80
  Male | 34 | 36 | 70
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 75 | 75 | 150

OUTCOME MEASURES:

1. Primary Outcome: Change in in Pain Score at 30 Minutes
Description: The primary outcome of this trial is the comparative change in participant's pain scores at 30 minutes post medication administration. Pain score is measured in a 11 point Likert Scale where 0 is no pain and 10 is extreme pain; 5 is moderate pain.
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IV SDK | K-BAN
Number analyzed (Participants) | 72 | 75
score on a scale | 4.7 (3.2) | 4.5 (2.8)

ADVERSE EVENTS:
Time Frame: 30 minutes
Arm/Group | IV SDK | K-BAN
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/75
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/75
Other Adverse Events (participants affected / at risk) | 0/75 | 0/75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-12): https://cdn.clinicaltrials.gov/large-docs/85/NCT04947085/Prot_SAP_002.pdf